CLINICAL TRIAL: NCT04640181
Title: A Phase 2-3, Multi-Center, Randomized Trial to Study the Potential Benefit of Factor Xa Inhibitor (Rivaroxaban) Versus Standard of Care Low Molecular Weight Heparin (Lovenox) in Hospitalized Patients With COVID-19 (XACT)
Brief Title: Factor Xa Inhibitor Versus Standard of Care Heparin in Hospitalized Patients With COVID-19 (XACT)
Acronym: XACT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: St. David's HealthCare (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-001708-41
Record Dates: First submitted 2020-11-19; First posted 2020-11-23 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Covid19
Keywords: Coronavirus; Enoxaparin; Rivaroxaban; Anticoagulants; Anti-inflammatory; Anti-viral; ARDS
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — Enoxaparin; Rivaroxaban

STUDY DESIGN:
Intervention Model Description: Open-label Multicenter Prospective Randomized Trial in hospitalized patients with severe acute respiratory syndrome (SARS)-CoV-2 infection. Patients will be randomized 1:1 to subcutaneous enoxaparin (Lovenox) versus rivaroxaban after hospitalization, with the exact dosing is based on an adaptive strategy.
Masking Description: Open label
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Adaptive Dosing: Enoxaparin (Active Comparator): * Low 40mg subcutaneous (SQ) daily, or
  * Intermediate 40mg SQ q12 hours, or
  * Therapeutic 1mg/kg SQ q12 hours
  Interventions: Drug: Enoxaparin
- Adaptive Dosing: Rivaroxaban (Active Comparator): * Low 10mg po daily
  * Intermediate 10mg po daily
  * Therapeutic 20mg po daily
  Interventions: Drug: Rivaroxaban

INTERVENTIONS:
Drug: Enoxaparin — Subcutaneous enoxaparin While hospitalized only.
  Arms: Adaptive Dosing: Enoxaparin
Drug: Rivaroxaban — Oral rivaroxaban While hospitalized and through discharge for a total of 28 days.
  Arms: Adaptive Dosing: Rivaroxaban

SUMMARY:
This study is a multicenter, randomized trial to study the potential benefit of treatments with a direct FXa inhibitor (rivaroxaban) versus standard of care dose subcutaneous low molecular weight heparin (LMWH) (Lovenox) in hospitalized subjects with COVID-19.

DETAILED DESCRIPTION:
As clinicians learn how to better care for hospitalized COVID-19 patients, the clinical picture of a hypercoagulable state with abnormal blood clotting has emerged. Fulminant heart, lung, kidney, and liver failure are hallmarks of COVID-19 non-survivors and have been associated with abnormal blood coagulation parameters, such as elevated D-Dimer levels. The current standard of care using prophylactic levels of subcutaneous heparin has not significantly mitigated the risk of patients entering a hypercoagulable state, however the dysregulated thrombotic and inflammatory events that drive poor outcomes in many COVID-19 patients may be amenable to early treatment with a factor Xa (FXa) inhibitor. The purpose of this study is to study the potential benefit of treatments with a direct FXa inhibitor (rivaroxaban) versus standard of care dose subcutaneous LMWH (Lovenox) in hospitalized subjects with COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 18-100 admitted to hospital with laboratory-confirmed SARS-CoV-2 infection
* Not be intubated or mechanically ventilated or imminently at risk for same or ICU admission within 24 hours of enrollment.
* Not be admitted for central nervous system (CNS) diagnosis
* Not have a current history of a condition requiring full therapeutic anticoagulation such as venous thromboembolism, atrial fibrillation.

Exclusion Criteria:

Medical Conditions

* Life expectancy of less than 6 months
* Active or recent gastrointestinal bleeding in the past 6 months
* Intracranial bleeding in the past 6 months
* Major trauma or head trauma in the past 2 months
* Major surgery in the past 2 months or planned within 2 weeks after completion of the study
* Recent spinal or epidural procedures in the past 2 weeks
* Ischemic stroke in the past 2 weeks
* History of intracranial neoplasm, arteriovenous malformation or aneurysm
* History of acquired or spontaneous impairment of hemostasis such as but not limited to hemophilia, idiopathic thrombocytopenic purpura (ITP), thrombotic thrombocytopenic purpura (TTP), von Willebrand disease
* Allergy to heparin or rivaroxaban or any factor Xa inhibitors, including a history of heparin-induced thrombocytopenia
* History of antiphospholipid syndrome
* End-stage renal failure requiring dialysis
* Valvular heart disease requiring chronic anticoagulation
* History of atrial fibrillation, atrial flutter or venous thromboembolic event (VTE) currently requiring anticoagulation
* History of solid organ transplant requiring immunosuppressant therapy
* Cancer requiring ongoing anticoagulation
* History of cirrhosis or liver failure, hepatorenal syndrome
* History of baseline bronchiectasis
* History of systemic lupus erythematosus or other autoimmune diseases requiring immunosuppressant therapy.

Vital signs

* Uncontrolled hypertension: systolic blood pressure (SBP) > 180 mm Hg or diastolic blood pressure (DBP) > 105mm Hg. Subjects who have a transient, higher blood pressure elevation (SBP 180-200 mm Hg) may enter the study if a repeat confirmation is back in range prior to enrollment.

Laboratory

* PT INR > 2.0.
* Platelet < 90 10^3/µL
* Total bilirubin > 3.0 mg/dL
* Hemoglobin < 9.0 g/dL
* Urine with gross hematuria (not due to menses)
* Estimated glomerular filtration rate (GFR) less than 30 mL/min calculated with the Cockcroft-Gault formula

Medications

* Patients on dual anti-platelet therapy
* Patients taking hypoxia-inducible factor prolyl hydroxylase inhibitors (such as roxadustat.)
* Erythropoiesis-stimulating agents (such as epoetin alfa, darbepoetin alfa)

Other COVID-19 drug studies or trials

* Any COVID19 vaccination trials
* Experimental COVID drug trial except for treatment(s) that has become accepted standard of care.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-06-28 (Actual); Study Completion 2021-06-28 (Actual)

PRIMARY OUTCOMES:
Death or 30-day all cause mortality | 30 days
Mechanical ventilation, intubation | 30 days
Transfer to an ICU setting | 30 days

SECONDARY OUTCOMES:
New requirement for hemodialysis (HD) or continuous renal replacement therapy (CRRT) or extracorporeal membrane oxygenation (ECMO) | 30 days
New thrombotic events | 30 days
Major bleeding event | 30 days
Time to recovery (defined as no limitation or minor limitation in activity level or hospitalized but require no oxygen) | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Edward Chafizadeh, MD, Principal Investigator — Cardio Texas, PLLC; Theresa Pham, MD, Principal Investigator — PPD Austin
Locations (1):
- St. David's Medical Center, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Drug information for Enoxaparin sodium provided by the National Library of Medicine — https://druginfo.nlm.nih.gov/drugportal/name/Enoxaparin+sodium
- See also: Xarelto (rivaroxaban) full prescribing information — http://www.janssenlabels.com/package-insert/product-monograph/prescribing-information/XARELTO-pi.pdf